CLINICAL TRIAL: NCT01590095
Title: WASH Benefits Bangladesh: A Cluster Randomized Controlled Trial of the Benefits of Water, Sanitation, Hygiene Plus Nutrition Interventions on Child Growth
Brief Title: WASH Benefits Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of California, Berkeley (Other); University of California, Davis (Other); Stanford University (Other); Emory University (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-11063; 2011-09-3652 (UC Berkeley)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-01

CONDITIONS: Malnutrition; Diarrhea; Child Development
Keywords: Chlorine water treatment; Point-of-use water treatment; Household water treatment with safe storage; Hand washing with soap; Hand hygiene; Latrines; Child potties; Point-of-use fortification; Lipid-based nutrient supplement; Environmental enteropathy; Tropical enteropathy; Gut function; Intestinal parasitic infection; Soil transmitted helminths; Intestinal protozoans; Antibody response; Water; Sanitation; Hand washing; Breast Feeding; Complementary Feeding; Micronutrients; Malnutrition; Nutrition Disorders; Diarrhea; Child Development
MeSH Terms: conditions — Malnutrition; Diarrhea; Sprue, Tropical; Intestinal Diseases, Parasitic; Breast Feeding; Nutrition Disorders | interventions — Water Quality; Sanitation; Hand Disinfection; Nutritional Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Water quality (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Water quality
- Sanitation (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Sanitation
- Hand washing (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Hand washing
- Combined WASH (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Water quality, Sanitation, Hand washing (Combined WASH)
- Nutrition (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Nutrition
- Nutrition + Combined WASH (Active Comparator): 90 clusters, approx. 720 newborns
  Interventions: Behavioral: Nutrition, Water quality, Sanitation, Hand washing
- Non-intervention (No Intervention): 180 clusters, approx. 1,440 newborns

INTERVENTIONS:
Behavioral: Water quality — Hardware: Free supplies chlorine tablets (Aquatabs; NaDCC) and a safe storage vessel to treat and store drinking water.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the treatment of all drinking water for children < 36 months of age.
  Arms: Water quality
Behavioral: Sanitation — Hardware: Free child potties, sani-scoop hoes to remove feces from household environments, latrine upgrades to a dual pit latrine Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the use of latrines for defecation and the removal of human and animal feces from the compound.
  Arms: Sanitation
Behavioral: Hand washing — Hardware: Hand washing stations, soapy water bottles located at hand washing locations, detergent soap to supply soapy water bottles.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on hand washing with soap at critical times around food preparation, defecation, and contact with feces.
  Arms: Hand washing
Behavioral: Water quality, Sanitation, Hand washing (Combined WASH) — Hardware: Free supplies Aquatabs; (NaDCC) and a safe storage vessel to treat and store drinking water. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the treatment of all drinking water for children < 36 months of age.
  Hardware: Free child potties, sani-scoop hoes to remove feces from household environments, latrine upgrades to a dual pit latrine. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on the use of latrines for defecation and the removal of human and animal feces from the compound.
  Hardware: Hand washing stations, soapy water bottles located at hand washing locations, detergent soap to supply soapy water bottles. Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages that focus on hand washing with soap at critical times around food preparation, defecation, and contact with feces.
  Arms: Combined WASH
Behavioral: Nutrition — Supplement: Lipid-based Nutrient Supplement (LNS) delivered daily from ages 6 to 24 months.
  Promotion: Local promoters will visit study compounds at least monthly to deliver behavior change messages modeled on those recommended in the Guiding Principles for Complementary Feeding of the Breastfed Child and the recent UNICEF Program Guide for Infant and Young Child Feeding Practices.General messages will include (1) practice exclusive breastfeeding from birth to 6 months of age and introduce complementary foods at 6 months of age while continuing to breastfeed; (2) continue breast feeding as you did before receiving LNS; (3) provide your child micronutrient-rich foods such as meat, fish, eggs, and vitamin A rich fruits and vegetables; and (4) feed your child at least 2-3 times per day when 6-8 months old and 3-4 times per day when 9-24 months old.
  Arms: Nutrition
Behavioral: Nutrition, Water quality, Sanitation, Hand washing — Each of the interventions described above for Water Quality, Sanitation & Hand washing (Combined WASH) Plus the intervention described above for nutrition.
  Arms: Nutrition + Combined WASH

SUMMARY:
Brief Summary:

The purpose of this study is to measure the independent and combined effects of interventions that improve water quality, sanitation, hand washing, and nutrition on child growth and development in the first years of life.

DETAILED DESCRIPTION:
Detailed Description:

Infection and inadequate diet are proximate risk factors for under-nutrition and early life growth faltering; the two processes likely act reciprocally in a vicious cycle that perpetuates physiologic and metabolic deficits and increases the risk of mortality. Children who exhibit growth faltering are more likely to have deficits in cognitive development and long-term human capital, and are more likely to have children who also suffer from growth deficits - perpetuating the cycle into the next generation.

There are two probable interdependent pathways that link enteric infections to child growth and development. The first pathway includes repeated infections the lead to acute illness or parasitic infection in the first years of life, which increase the risk of stunting and subsequent cognitive deficits in childhood and later in life. The second pathway is through a subclinical condition called environmental enteropathy (EE).

There is limited evidence to demonstrate whether or not water quality, sanitation, and hand washing (WASH) interventions can improve measures of EE, child growth and development, and whether nutritional interventions could be enhanced if provided concurrently with WASH interventions. To help fill this evidence gap, the WASH Benefits study will deliver randomized interventions designed to reduce infection and improve nutrition, and will measure intervention effects on child illness, growth and development. WASH Benefits includes two, comparable but standalone trials in Bangladesh and Kenya that are registered under separate protocols.

In Bangladesh, the study will include 720 clusters, and each cluster will enroll 8 household compounds (baris) with pregnant women in their second or third trimester. The study will randomize 90 clusters to each of 6 active intervention arms (water quality, sanitation, hand washing, combined WSH, nutrition, nutrition+WSH), and 180 clusters to a standard practices non-intervention arm. Children born into the cohort will be followed for 2 years after the intervention, with measurements at 12 and 24 months after intervention delivery. (anticipated age range: 20 - 27 months old at the final measurement). At the 12- and 24-month follow-up visits, the study will collect child anthropometric measurements and caregiver-reported diarrhea. In the final visit the study will administer a test to measure child development outcomes. The study will collect urine, blood, and stool specimens from a subsample of 1,500 children distributed across four arms of the study (Control, combined WSH, Nutrition, Nutrition+WSH) to measure biomarkers of gut function and intestinal parasitic infections at the 12- and 24-month follow-up visits. In addition, the study will collect specimens (blood, stool) from children 18 - 27 months old at baseline who are living in the same compound as target children to test for intestinal parasitic infections. At 24-months in all arms, the study will collect specimens stool from target children, children 18 - 27 months old at baseline, a school-aged child, and an adult who are living in the same compound as target children to test for intestinal parasitic infections. At 36-months in all arms, the study will collect specimens stool from target children, a school-aged child, and an adult who are living in the same compound as target children to test for intestinal parasitic infections.

ELIGIBILITY:
Inclusion Criteria:

(1) Infants (target child) will be eligible to participate in the study if they are:

1. They are in utero at the baseline survey
2. Their parents/guardians are planning to stay in the study village for the next 12 months (if a mother is planning to give birth at her natal home and then return, she will still be a candidate for enrollment)

(2) Children < 36 months old at baseline that are living in the compound of a target child will be eligible to participate in diarrhea measurement if:

1. They are < 36 months old at the baseline survey
2. Their parents/guardians are planning to stay in the study village for the next 12 months

(3) Children 18 - 27 months old at baseline that are living in the compound of a target child will be eligible to participate in intestinal parasite specimen collection if:

1. They are 18 - 27 months old at the baseline survey
2. Their parents/guardians are planning to stay in the study village for the next 12 months

Ages: 1 Day to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5040 (Estimated)
Dates: Start 2012-05; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Length-for-Age Z-scores | Measured 24 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 24monthsafter intervention. Measurement techniques follow the FANTA 2003 protocol.
Diarrhea Prevalence Diarrhea Prevalence Diarrhea Prevalence Diarrhea Prevalence | Measured 12- and 24-months after intervention
  Diarrhea is defined as 3+ loose or watery stools in 24 hours or 1+ stools with blood in 24 hours. Diarrhea will be measured in interviews using caregiver-reported symptoms with 2-day and 7-day recall, measured 12- and 24-monthsafter intervention.

SECONDARY OUTCOMES:
Length-for-Age Z-scores | Measured 12 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 12monthsafter intervention. Measurement techniques follow the FANTA 2003 protocol.
Stunting Prevalence | Measured 24 months after intervention
  Child's recumbent length, standardized to Z-scores using the WHO 2006 growth standards, measured 24monthsafter intervention. Measurement techniques follow the FANTA 2003 protocol. Children with length-for-age Z-scores < - 2 will be classified as stunted.
Enteropathy Biomarkers | Measured 12- and 24 months after intervention
  The lactulose / mannitol dual sugar permeability test will be administered to children. The ratio of the recovery of the two sugars in the urine will be used to calculate the L:M ratio, and we will compare groups using logged values of the ratio. We will additionally measure Total IgG antibody titers in the blood, and we will compare groups using logged values of the antibody levels.
ASQ Child Development Scores | Measured 24 months after intervention
  Interviewers will administer a locally adapted version of the Ages and Stages Questionnaire (ASQ)to children after 24 months of intervention. The ASQ includes item sets of caregiver-reported milestones that measure child development in three separate domains (gross motor, communication, personal/social skills).

OTHER OUTCOMES:
Infection with ascaris, trichuris, hookworm, and giardia | Measured 24 months after interventions began
  Infection with soil transmitted helminths (ascaris, trichuris, hookworm) will be enumerated in stool collected from all index children and one older child per study compound. Giardia will also be measured in stool samples collected from these children. Prevalence and eggs per gram of feces will be recorded.
Hemoglobin concentration and anemia | Measured 24 months after interventions began
  Hemoglobin concentrations will be measured using venous blood samples with a Hemocue 301 analyzer
Micronutrient status, including iron, vitamin A, folate, and B12 | Measured 24 months after interventions began
  Iron status will be assessed using the biomarkers of ferritin, soluble transferrin receptor (sTfR), and hepcidin. Vitamin A status will be assessed using retinol binding protein. Folate and B12 status will be measured using plasma folate and B12.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Luby, MD, Principal Investigator — Stanford University
Locations (1):
- Dr. Mahbubur Rahman, Dhaka, Bangladesh

REFERENCES:
- [Derived] Chen B, Mertens AN, Lin CH, Tan ST, Jamshed F, Figueroa D, Hemlock C, Butzin-Dozier Z, Fernald LC, Stewart CP, Hubbard AE, Rahman MZ, Ali S, Arnold BF, Dhabhar FS, Granger DA, Rahman M, Luby SP, Colford JM Jr, Lin A. Associations Between Micronutrient Status, Hormones, and Immune Status During Pregnancy and Child Growth in Rural Bangladesh: A Prospective Cohort Study. Curr Dev Nutr. 2025 Nov 8;9(12):107596. doi: 10.1016/j.cdnut.2025.107596. eCollection 2025 Dec. PMID 41467215
- [Derived] Tofail F, Pitchik HO, Islam M, Khan R, Shoab AK, Akter F, Aktar S, Huda TMN, Rahman M, Winch PJ, Luby SP, Fernald LCH. Effects of early water, sanitation, handwashing, and nutrition interventions on child development at school age: a follow-on study of a cluster-randomized trial in rural Bangladesh. PLoS Med. 2025 Dec 16;22(12):e1004793. doi: 10.1371/journal.pmed.1004793. eCollection 2025 Dec. PMID 41401135
- [Derived] Lin A, Mertens AN, Rahman MZ, Tan ST, Il'yasova D, Spasojevic I, Ali S, Stewart CP, Fernald LCH, Kim L, Yan L, Meyer A, Karim MR, Shahriar S, Shuman G, Arnold BF, Hubbard AE, Famida SL, Akther S, Hossen MS, Mutsuddi P, Shoab AK, Shalev I, Rahman M, Unicomb L, Heaney CD, Kariger P, Colford JM Jr, Luby SP, Granger DA. A cluster-randomized trial of water, sanitation, handwashing and nutritional interventions on stress and epigenetic programming. Nat Commun. 2024 Apr 26;15(1):3572. doi: 10.1038/s41467-024-47896-z. PMID 38670986
- [Derived] Contreras JD, Islam M, Mertens A, Pickering AJ, Arnold BF, Benjamin-Chung J, Hubbard AE, Rahman M, Unicomb L, Luby SP, Colford JM Jr, Ercumen A. Evaluation of an on-site sanitation intervention against childhood diarrhea and acute respiratory infection 1 to 3.5 years after implementation: Extended follow-up of a cluster-randomized controlled trial in rural Bangladesh. PLoS Med. 2022 Aug 8;19(8):e1004041. doi: 10.1371/journal.pmed.1004041. eCollection 2022 Aug. PMID 35939520
- [Derived] Lin A, Mertens AN, Arnold BF, Tan S, Lin J, Stewart CP, Hubbard AE, Ali S, Benjamin-Chung J, Shoab AK, Rahman MZ, Famida SL, Hossen MS, Mutsuddi P, Akther S, Rahman M, Unicomb L, Naved RT, Mamun MMA, Parvin K, Dhabhar FS, Kariger P, Fernald LC, Luby SP, Colford JM Jr. Telomere length is associated with growth in children in rural Bangladesh. Elife. 2021 Sep 8;10:e60389. doi: 10.7554/eLife.60389. PMID 34494545
- [Derived] Kwong LH, Sen D, Islam S, Shahriar S, Benjamin-Chung J, Arnold BF, Hubbard A, Parvez SM, Islam M, Unicomb L, Rahman MM, Nelson K, Colford JM Jr, Luby SP, Ercumen A. Effect of sanitation improvements on soil-transmitted helminth eggs in courtyard soil from rural Bangladesh: Evidence from a cluster-randomized controlled trial. PLoS Negl Trop Dis. 2021 Jul 28;15(7):e0008815. doi: 10.1371/journal.pntd.0008815. eCollection 2021 Jul. PMID 34319986
- [Derived] Contreras JD, Islam M, Mertens A, Pickering AJ, Kwong LH, Arnold BF, Benjamin-Chung J, Hubbard AE, Alam M, Sen D, Islam S, Rahman M, Unicomb L, Luby SP, Colford JM, Ercumen A. Longitudinal Effects of a Sanitation Intervention on Environmental Fecal Contamination in a Cluster-Randomized Controlled Trial in Rural Bangladesh. Environ Sci Technol. 2021 Jun 15;55(12):8169-8179. doi: 10.1021/acs.est.1c01114. Epub 2021 Jun 4. PMID 34086447
- [Derived] Parvez SM, Rahman MJ, Azad R, Rahman M, Unicomb L, Ashraf S, Mondol MH, Jahan F, Winch PJ, Luby SP. Achieving equitable uptake of handwashing and sanitation by addressing both supply and demand-based constraints: findings from a randomized controlled trial in rural Bangladesh. Int J Equity Health. 2021 Jan 6;20(1):16. doi: 10.1186/s12939-020-01353-7. PMID 33407549
- [Derived] Ercumen A, Benjamin-Chung J, Arnold BF, Lin A, Hubbard AE, Stewart C, Rahman Z, Parvez SM, Unicomb L, Rahman M, Haque R, Colford JM Jr, Luby SP. Effects of water, sanitation, handwashing and nutritional interventions on soil-transmitted helminth infections in young children: A cluster-randomized controlled trial in rural Bangladesh. PLoS Negl Trop Dis. 2019 May 3;13(5):e0007323. doi: 10.1371/journal.pntd.0007323. eCollection 2019 May. PMID 31050672
- [Derived] Lin A, Ali S, Arnold BF, Rahman MZ, Alauddin M, Grembi J, Mertens AN, Famida SL, Akther S, Hossen MS, Mutsuddi P, Shoab AK, Hussain Z, Rahman M, Unicomb L, Ashraf S, Naser AM, Parvez SM, Ercumen A, Benjamin-Chung J, Haque R, Ahmed T, Hossain MI, Choudhury N, Jannat K, Alauddin ST, Minchala SG, Cekovic R, Hubbard AE, Stewart CP, Dewey KG, Colford JM, Luby SP. Effects of Water, Sanitation, Handwashing, and Nutritional Interventions on Environmental Enteric Dysfunction in Young Children: A Cluster-randomized, Controlled Trial in Rural Bangladesh. Clin Infect Dis. 2020 Feb 14;70(5):738-747. doi: 10.1093/cid/ciz291. PMID 30963177
- [Derived] Stewart CP, Dewey KG, Lin A, Pickering AJ, Byrd KA, Jannat K, Ali S, Rao G, Dentz HN, Kiprotich M, Arnold CD, Arnold BF, Allen LH, Shahab-Ferdows S, Ercumen A, Grembi JA, Naser AM, Rahman M, Unicomb L, Colford JM Jr, Luby SP, Null C. Effects of lipid-based nutrient supplements and infant and young child feeding counseling with or without improved water, sanitation, and hygiene (WASH) on anemia and micronutrient status: results from 2 cluster-randomized trials in Kenya and Bangladesh. Am J Clin Nutr. 2019 Jan 1;109(1):148-164. doi: 10.1093/ajcn/nqy239. PMID 30624600
- [Derived] Parvez SM, Azad R, Rahman M, Unicomb L, Ram PK, Naser AM, Stewart CP, Jannat K, Rahman MJ, Leontsini E, Winch PJ, Luby SP. Achieving optimal technology and behavioral uptake of single and combined interventions of water, sanitation hygiene and nutrition, in an efficacy trial (WASH benefits) in rural Bangladesh. Trials. 2018 Jul 6;19(1):358. doi: 10.1186/s13063-018-2710-8. PMID 29976251
- [Derived] Rahman M, Ashraf S, Unicomb L, Mainuddin AKM, Parvez SM, Begum F, Das KK, Naser AM, Hussain F, Clasen T, Luby SP, Leontsini E, Winch PJ. WASH Benefits Bangladesh trial: system for monitoring coverage and quality in an efficacy trial. Trials. 2018 Jul 6;19(1):360. doi: 10.1186/s13063-018-2708-2. PMID 29976234
- [Derived] Lin A, Ercumen A, Benjamin-Chung J, Arnold BF, Das S, Haque R, Ashraf S, Parvez SM, Unicomb L, Rahman M, Hubbard AE, Stewart CP, Colford JM Jr, Luby SP. Effects of Water, Sanitation, Handwashing, and Nutritional Interventions on Child Enteric Protozoan Infections in Rural Bangladesh: A Cluster-Randomized Controlled Trial. Clin Infect Dis. 2018 Oct 30;67(10):1515-1522. doi: 10.1093/cid/ciy320. PMID 29669039
- [Derived] Tofail F, Fernald LC, Das KK, Rahman M, Ahmed T, Jannat KK, Unicomb L, Arnold BF, Ashraf S, Winch PJ, Kariger P, Stewart CP, Colford JM Jr, Luby SP. Effect of water quality, sanitation, hand washing, and nutritional interventions on child development in rural Bangladesh (WASH Benefits Bangladesh): a cluster-randomised controlled trial. Lancet Child Adolesc Health. 2018 Apr;2(4):255-268. doi: 10.1016/S2352-4642(18)30031-2. PMID 29616235
- [Derived] Lin A, Arnold BF, Mertens AN, Lin J, Benjamin-Chung J, Ali S, Hubbard AE, Stewart CP, Shoab AK, Rahman MZ, Hossen MS, Mutsuddi P, Famida SL, Akther S, Rahman M, Unicomb L, Dhabhar FS, Fernald LCH, Colford JM Jnr, Luby SP. Effects of water, sanitation, handwashing, and nutritional interventions on telomere length among children in a cluster-randomized controlled trial in rural Bangladesh. Elife. 2017 Oct 5;6:e29365. doi: 10.7554/eLife.29365. PMID 28980942
- [Derived] Arnold BF, Null C, Luby SP, Unicomb L, Stewart CP, Dewey KG, Ahmed T, Ashraf S, Christensen G, Clasen T, Dentz HN, Fernald LC, Haque R, Hubbard AE, Kariger P, Leontsini E, Lin A, Njenga SM, Pickering AJ, Ram PK, Tofail F, Winch PJ, Colford JM Jr. Cluster-randomised controlled trials of individual and combined water, sanitation, hygiene and nutritional interventions in rural Bangladesh and Kenya: the WASH Benefits study design and rationale. BMJ Open. 2013 Aug 30;3(8):e003476. doi: 10.1136/bmjopen-2013-003476. PMID 23996605
- See also: Related protocol — http://clinicaltrials.gov/ct2/show/NCT01704105
- See also: Click here for more informaiton about the study — http://www.washbenefits.net